CLINICAL TRIAL: NCT02483338
Title: Does the FASS (Facial Action Summary Score) Scale Allow to Differentiate the Pain of Postoperative Anxiety in Children Under 7 Years?
Brief Title: FASS (Facial Action Summary Score) Scale to Differentiate the Pain of Postoperative Anxiety in Children Under 7 Years
Acronym: FASS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 8824; 2011-A00533-38 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2015-06-24; First posted 2015-06-26 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-06

CONDITIONS: Postoperative Pain
Keywords: Psychometric validity; Pain scale; Postoperative; Children
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Children surgery (Other)
  Interventions: Behavioral: Assessment of pain

INTERVENTIONS:
Behavioral: Assessment of pain — Assessment of pain using FASS but without using this score to manage pain

SUMMARY:
This study aims to evaluate the psychometric validity of FASS (Facial Summary Score Scale) to assess postoperative children pain.

ELIGIBILITY:
Inclusion Criteria:

* Children surgery
* Younger than 7 years old
* Elective surgery
* Patient whose parents will have given their non-opposition

Exclusion Criteria:

* Psychological retardation
* Chronic pain

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2011-07; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
FASS (Facial Action Summary Score) | As soon as the child arrive in recovery room or / and the extubation, before and after the administration of analgesics

CONTACTS AND LOCATIONS:
Overall Officials: Sophie SB BRINGUIER, HP, Principal Investigator — Department of Anesthesia Resuscitation at the Hospital Lapeyronie in Montpellier
Locations (1):
- University hospital Lapeyronie, Montpellier, France